CLINICAL TRIAL: NCT02758509
Title: Efficacy and Safety of Interferon Based Therapy and Interferon-free Direct-acting Antivirals in Cirrhotic Patients With Hepatitis C. Impact of Antiviral Therapy on Gastroesophageal Varices.
Brief Title: Impact of Antiviral Therapy on Gastroesophageal Varices.
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, José Antonio Carrion, PhD, Parc de Salut Mar
Other Study IDs: PROGRESSIVE-C
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Chronic Hepatitis C; Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis | interventions — peginterferon alfa-2a; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; ledipasvir, sofosbuvir drug combination; Viekira Pak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PEG/RBV: Pegylated interferon alfa-2a 180 microg/week plus ribavirin 800-1200 mg during 48 weeks according to routine practice and European Guidelines (EASL recommendations 2011)
  Interventions: Drug: Pegylated interferon alfa-2a + Ribavirin
- PEG/RBV+BOC or TVR: Boceprevir 800 mg/8h or Telaprevir 750 mg/8h plus Pegylated interferon alfa-2a 180 microg/week plus ribavirin 800-1200 mg during 48 weeks according to routine practice and European Guidelines (EASL recommendations 2014)
  Interventions: Drug: Pegylated interferon alfa-2a + Ribavirin + Boceprevir; Drug: Pegylated interferon alfa-2a + Ribavirin +Telaprevir
- IF-DAAs: Interferon-free direct-acting antiviral combinations according to routine practice and European Guidelines (EASL recommendations 2015)
  * Fixed-dose combination of sofosbuvir (400 mg) and ledipasvir (90 mg) daily +/- ribavirin 12-24 weeks
  * Fixed-dose combination of ombitasvir (75 mg), paritaprevir (12.5 mg) and ritonavir (50 mg) in one single tablet (two tablets once daily) and dasabuvir (250 mg) (one tablet twice daily) with ribavirin 800-1200 mg 12 weeks (Genotype 1b) or 24 weeks (genotype 1a)
  * Daily sofosbuvir (400 mg) and daily simeprevir (150 mg) +/- ribavirin 12-24 weeks
  * Daily sofosbuvir (400 mg) and daily daclatasvir (60 mg) +/- ribavirin 12-24 weeks
  Interventions: Drug: Ledipasvir/Sofosbuvir; Drug: Ombitasvir/paritaprevir/ritonavir+Dasabuvir; Drug: Daclatasvir+Sofosbuvir; Drug: Simeprevir+Sofosbuvir

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a + Ribavirin
  Groups: PEG/RBV
Drug: Pegylated interferon alfa-2a + Ribavirin + Boceprevir
  Groups: PEG/RBV+BOC or TVR
Drug: Pegylated interferon alfa-2a + Ribavirin +Telaprevir
  Groups: PEG/RBV+BOC or TVR
Drug: Ledipasvir/Sofosbuvir
  Groups: IF-DAAs
Drug: Ombitasvir/paritaprevir/ritonavir+Dasabuvir
  Groups: IF-DAAs
Drug: Daclatasvir+Sofosbuvir
  Groups: IF-DAAs
Drug: Simeprevir+Sofosbuvir
  Groups: IF-DAAs

SUMMARY:
Hepatitis C virus (HCV) chronic infection affects 200 million people worldwide. HCV antiviral treatment has evolved rapidly since 2011. The use of pegylated interferon (PEG-INF) with ribavirin (RBV) has supposed high serious adverse events (SAEs) and low efficacy, especially in patients with cirrhosis. The introduction of 1st generation protease inhibitors (PIs) in genotype-1 (GT1) HCV, such as boceprevir (BOC) and telaprevir (TVR), improved the efficacy but increased the SAEs. Currently, interferon-free direct-acting antivirals (IF-DAAs) achieve great effectiveness with minimum SAEs. However, studies evaluating efficacy and safety of DAAs in cirrhotic patients are limited in real clinical practice. The aim of our study is to evaluate in HCV-cirrhotic patients the efficacy and safety of 3 treatment strategies (PEG-IFN/RBV, PEG-IFN/RBV/PIs, and IF-DAAs) in routine practice according to European guidelines from 2010 to 2015. The secondary aim is to evaluate the impact of sustained virological response on gastroesophageal varices (GOV).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Signed informed consent.
* Chronic hepatitis C (anti-HCV antibodies and detectable HCV-RNA).
* Liver cirrhosis (transient elastography ≥ 14 kPa).
* Baseline upper gastrointestinal endoscopy to assess gastroesophageal varices

Exclusion Criteria:

* Negative to provide signed informed consent.
* Negative to perform gastrointestinal endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C by genotype 1 and liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2010-01-01; Primary Completion 2017-06-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
sustained virological response (SVR) | 12 weeks after treatment completion
  undetectable HCV viral load 12 weeks after the end of antiviral treatment in each cohort of antiviral treatment

SECONDARY OUTCOMES:
Number of patients with gastroesophageal varices | gastroesophageal varices (GOV) before antiviral treatment and 12-24 weeks after treatment completion
  Number of patients with GOV before and 12-24 weeks after treatment completion in patients with or without SVR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puigvehi M, Londono MC, Torras X, Lorente S, Vergara M, Morillas RM, Masnou H, Serrano T, Miquel M, Gallego A, Lens S, Carrion JA. Impact of sustained virological response with DAAs on gastroesophageal varices and Baveno criteria in HCV-cirrhotic patients. J Gastroenterol. 2020 Feb;55(2):205-216. doi: 10.1007/s00535-019-01619-0. Epub 2019 Sep 6. PMID 31493238